CLINICAL TRIAL: NCT04322331
Title: The Different Transcriptional Characterization Of The Tumor Immune Microenvironment of Luminal A Breast Cancer With Different Lymph Node Metastasas Status
Brief Title: Tumor Immune Mechanism of Axillary Lymph Node Metastasis in Early Luminal Type A Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IO Panel
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Immune Microenvironment; Luminal A; Lymph Node Metastases
MeSH Terms: conditions — Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T1N+: T1 tumor with positive lymph node,N1/N2/N3
  Interventions: Other: no intervention
- T2/T3N0: T2/T3 tumor with negative lymph node
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Luminal type A breast cancer is a type with good clinical prognosis, and the proportion of lymph node metastasis is low, but a small number of patients have more lymph node metastasis when the primary tumor is very small, and the survival is poor, suggesting that this part of Luminal A breast cancer has the different expression of some genes from that of general Luminal A breast cancer, which affects tumor invasion and participates in the occurrence of tumor metastasis. But the mechanism is not clear, especially in the current tumor microenvironment and immune related mechanisms.We want to investigated the relationship of the transcriptional tumor immune microenvironment with early lymph node metastasis among Luminal A type breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* invasive breast cancer with Luminal A type;T1 with positive lymph node or T2/T3 with negative lymph node

Exclusion Criteria:

* Missing specimen

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: invasive breast cancer patients with Luminal A type. Stage T1N1/T1N2/T1N3 are in group 1; stage T2N0/T3N0 are in group 2
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Transcriptional Characterization | 2020-12
  the relationship of the transcriptional tumor immune microenvironment with lymph node metastases in Luminal A breast tumor;Differences in RNA copy numbers of different genes （using IO Panel） between the two groups of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Peking university people's hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol